CLINICAL TRIAL: NCT00303784
Title: A Randomized-Controlled Trial of Transcutaneous Oestrogen Patches Versus LHRH Agonists in Prostate Cancer
Brief Title: Prostate Adenocarcinoma TransCutaneous Hormones
Acronym: PATCH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000455583; MRC-PATCH (Other Grant/Funding Number: MRC); EU-205106 (Other: EU); MRC-PR09 (Other: MRC); ISRCTN70406718 (Registry Identifier: ISRCTN70406718); 2005-001030-33 (EudraCT Number)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Anemia; Cardiovascular Complications; Hot Flashes; Osteoporosis; Prostate Cancer
Keywords: hot flashes; anemia; osteoporosis; cardiovascular complications; recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Anemia; Hot Flashes; Osteoporosis; Prostatic Neoplasms | interventions — Goserelin; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LHRH agonists (Active Comparator): Patients randomised to the control arm will receive continuous treatment with LHRH agonists as per local practice. Treatment should continue for at least 3 years. LHRH antagonists, such as degarelix, are not allowed on the trial. The recommended "anti-flare" medication is bicalutamide and should be prescribed according to local practice. Control arm medication should be obtained from the hospital pharmacy or GP as per local practice.
  Interventions: Drug: Goserelin
- Oestrogen Patches (Experimental): Patients randomised to the investigational arm will receive transcutaneous oestrogen patches (100 micrograms/24 hours). Treatment should be planned to continue for at least 3 years. For patients prescribed bicalutamide or flutamide prior to randomisation, this treatment should be discontinued before treatment with the patches can commence (no washout period is needed).
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Goserelin — 3.6mg implant, in pre-filled syringe
  Other Names: Zoladex
  Arms: LHRH agonists
Drug: Estradiol — Each patch contains 3 mg of estradiol hemihydrate in a patch size of 30 cm2, releasing 100 micrograms of estradiol per 24 hours.
  Other Names: FemSeven
  Arms: Oestrogen Patches

SUMMARY:
RATIONALE: The increasingly prolonged and extended use of androgen deprivation therapy (ADT) in the treatment of prostate cancer, usually achieved through the administration of LHRH agonists, has raised concerns about long-term toxicities, in particular osteoporosis and adverse metabolic changes which may be associated with type II diabetes and increased cardiovascular risk. An alternative approach is to investigate other methods of ADT. Oral oestrogen has been shown to be as effective as LHRH and surgical orchidectomy in achieving castrate levels of testosterone and has equivalent or improved prostate cancer outcomes but is not used routinely as first-line therapy because of the risk of cardiovascular system (CVS) complications. The CVS complications have been attributed to first-pass hepatic metabolism. Administering oestrogen parenterally avoids the entero-hepatic circulation and so is expected to mitigate the risk of CVS toxicity whilst still effectively suppressing testosterone to castrate levels. This hypothesis has been supported by results from the early stages of this trial which have provided sufficient indication of the safety and efficacy of the patches to warrant further investigation of the treatment in this setting, as recommended by the IDMC..

PURPOSE: This randomized phase III trial is studying how well the estrogen skin patch works compared with luteinizing hormone-releasing hormone agonist injections in treating patients with locally advanced or metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival and overall survival of patients with locally advanced or metastatic prostate cancer treated with transcutaneous estrogen patches vs luteinizing hormone-releasing hormone analogues.

Secondary

* Compare the cardiovascular system-related morbidity and mortality in patients treated with these regimens
* Compare the activity of these treatments, in terms of castrate level of hormones, failure-free survival, and biochemical failure, in these patients.
* Compare other toxicities, including osteoporosis, hot flushes, gynecomastia, and anemia, in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms at 1(control):1 (patch) ratio.

* Arm I (control): Patients receive luteinizing hormone-releasing hormone agonists as per local practice in the absence of unacceptable toxicity.
* Arm II (patch): Patients receive 4 transcutaneous estrogen patches, changing twice weekly for 4 weeks. Patients' testosterone levels are measured at week 4. Patients whose testosterone level is > 1.7 nmol/L continue to receive patch as before and have their testosterone level measured every 2 weeks. Patients whose testosterone level is < 1.7 nmol/L at week 4 or any other point receive 3 transcutaneous estrogen patches changed twice weekly in the absence of unacceptable toxicity.

Quality of life is assessed at baseline; at weeks 4, 8, and 12; every 3 months for 24 months.

After completion of study treatment, patients are followed periodically.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 2200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must meet 1 of the following criteria:

  * Newly diagnosed patients with any of the following:

    * Stage T3 or T4, NX, M0 histologically confirmed prostate adenocarcinoma with prostate-specific antigen (PSA) ≥ 20 ng/mL or Gleason score ≥ 6
    * Any T, N+, M0, or any T, any N, M+ histologically confirmed prostate adenocarcinoma
    * Multiple sclerotic bone metastases with a PSA ≥ 50 ng/mL without histological confirmation
  * Patients with histologically confirmed prostate adenocarcinoma previously treated with radical surgery or radiotherapy who are currently in relapse with on of the following:

    * PSA ≥ 4 ng/mL and rising with doubling time less than 6 months
    * PSA ≥ 20 ng/mL
* Must have written informed consent
* Intention to treat with long-term androgen-deprivation therapy
* Normal testosterone level prior to hormonal treatment

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* No other prior or current malignant disease or cardiovascular system disease that is likely to interfere with study treatment or assessment
* No cardiovascular disease, including any of the following:

  * History of cerebral ischemia (e.g., stroke or transient ischemic attack) within the past 2 years
  * History of deep vein thrombosis or pulmonary embolism confirmed radiologically
  * History of myocardial infarction (MI) within the past 6 months OR MI more than 6 months ago with evidence of q-wave anterior infarct on ECG

    * ECHO or MUGA required for patients with history of ischemic heart disease
  * Left Ventricular Ejection Fraction ≤ 40%
* No condition or situation that could preclude protocol treatment or compliance with follow-up schedule

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 12 months since prior adjuvant or neoadjuvant hormonal therapy for localized prostate cancer AND therapy lasted ≤ 12 months in duration
* No prior systemic therapy for locally advanced or metastatic prostate cancer
* No concurrent participation in another clinical trial of prostate cancer treatment that would preclude study therapy or outcome measures
* Concurrent prophylactic radiotherapy to prevent gynecomastia allowed

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2006-03 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Up to 180 months
Overall Survival | Up to 180 months

SECONDARY OUTCOMES:
Hormone activity by castrate levels of hormones | Up to 180 months
Other toxicity | Up to 180 months
Cardiovascular morbidity | Up to 180 months
Cardiovascular mortality | Up to 180 months
Quality of Life | Up to 24 months
  will be measured using patient-completed questionnaires, EORTC QLQ-C30 and PR25 which is prostate specific

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Abel, Study Chair — Charing Cross Hospital
Locations (32):
- United Kingdom (32):
  - Queen's Hospital, Burton-on-Trent, England
  - Addenbrooke's Hospital, Cambridge, England
  - Walsgrave Hospital, Coventry, England
  - Mid Cheshire Hospitals Trust- Leighton Hopsital, Crewe, England
  - Mayday University Hospital, Croydon, England
  - Derbyshire Royal Infirmary, Derby, England
  - Castle Hill Hospital, East Yorkshire, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Grantham and District Hospital, Grantham, Lincolnshire, England
  - Ipswich Hospital, Ipswich, England
  - Kidderminster Hospital, Kidderminster Worcestershire, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - St. Mary's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Maidstone Hospital, Maidstone, England
  - James Cook University Hospital, Middlesbrough, England
  - Nottingham City Hospital, Nottingham, England
  - Kings Mill Hospital, Nottinghamshire, England
  - George Eliot Hospital, Nuneaton, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - Hope Hospital, Salford, England
  - Scarborough General Hospital, Scarborough, England
  - Stepping Hill Hospital, Stockport, England
  - Hillingdon Hospital, Uxbridge, England
  - Walsall Manor Hospital, Walsall, England
  - Warwick Hospital, Warwick, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil, England
  - Ayr Hospital, Ayr, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Derived] Gilbert DC, Nankivell M, Rush H, Clarke NW, Mangar S, Al-Hasso A, Rosen S, Kockelbergh R, Sundaram SK, Dixit S, Laniado M, McPhail N, Shaheen A, Brown S, Gale J, Deighan J, Marshall J, Duong T, Macnair A, Griffiths A, Amos CL, Sydes MR, James ND, Parmar MKB, Langley RE. A Repurposing Programme Evaluating Transdermal Oestradiol Patches for the Treatment of Prostate Cancer Within the PATCH and STAMPEDE Trials: Current Results and Adapting Trial Design. Clin Oncol (R Coll Radiol). 2024 Jan;36(1):e11-e19. doi: 10.1016/j.clon.2023.10.054. Epub 2023 Nov 8. PMID 37973477
- [Derived] Gilbert DC, Duong T, Sydes M, Bara A, Clarke N, Abel P, James N, Langley R, Parmar M; STAMPEDE and PATCH Trial Management Groups. Transdermal oestradiol as a method of androgen suppression for prostate cancer within the STAMPEDE trial platform. BJU Int. 2018 May;121(5):680-683. doi: 10.1111/bju.14153. Epub 2018 Feb 28. No abstract available. PMID 29388336
- [Derived] Langley RE, Kynaston HG, Alhasso AA, Duong T, Paez EM, Jovic G, Scrase CD, Robertson A, Cafferty F, Welland A, Carpenter R, Honeyfield L, Abel RL, Stone M, Parmar MK, Abel PD. A Randomised Comparison Evaluating Changes in Bone Mineral Density in Advanced Prostate Cancer: Luteinising Hormone-releasing Hormone Agonists Versus Transdermal Oestradiol. Eur Urol. 2016 Jun;69(6):1016-25. doi: 10.1016/j.eururo.2015.11.030. Epub 2015 Dec 17. PMID 26707868
- [Derived] Langley RE, Cafferty FH, Alhasso AA, Rosen SD, Sundaram SK, Freeman SC, Pollock P, Jinks RC, Godsland IF, Kockelbergh R, Clarke NW, Kynaston HG, Parmar MK, Abel PD. Cardiovascular outcomes in patients with locally advanced and metastatic prostate cancer treated with luteinising-hormone-releasing-hormone agonists or transdermal oestrogen: the randomised, phase 2 MRC PATCH trial (PR09). Lancet Oncol. 2013 Apr;14(4):306-16. doi: 10.1016/S1470-2045(13)70025-1. Epub 2013 Mar 4. PMID 23465742
- See also: Study homepage at the MRC CTU at UCL — http://www.ctu.mrc.ac.uk/our_research/research_areas/cancer/studies/patch_pr09/